CLINICAL TRIAL: NCT00791765
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Etanercept in Treating Scalp Involvement in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Moderate to Severe Plaque Psoriasis With Scalp Involvement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20080014
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Psoriasis
Keywords: Scalp; Psoriasis; Plaque Psoriasis; Skin Diseases; Moderate to severe plaque psoriasis; etanercept
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo BIW/Etanercept 50 mg BIW (Experimental): Participants received placebo subcutaneous injections twice per week (BIW) for the first 12 weeks of the study. From Week 12 to Week 24, participants received etanercept 50 mg BIW.
  Interventions: Biological: Etanercept; Biological: Placebo
- Etanercept 50 mg BIW/Etanercept 50 mg QW (Experimental): Participants received etanercept 50 mg by subcutaneous injection twice per week (BIW) for the first 12 weeks of the study. From Week 12 to Week 24, participants received etanercept 50 mg once per week (QW) and placebo once per week.
  Interventions: Biological: Etanercept; Biological: Placebo

INTERVENTIONS:
Biological: Etanercept — Etanercept for subcutaneous injection.
  Other Names: Enbrel®
Biological: Placebo — Placebo for subcutaneous injection.

SUMMARY:
The purpose of this study is to determine if etanercept is effective in the treatment of scalp involvement in moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent before any study-specific procedure
* Be male or female greater than or equal to 18 years of age at time of screening
* Has stable moderate to severe plaque psoriasis for at least 6 months
* Affected body surface area (BSA) greater than or equal to 10%
* Psoriasis Area and Severity Index (PASI) score greater than or equal to 10
* At least 30 percent affected scalp surface area
* Psoriasis Scalp Severity Index (PSSI) score greater than or equal to 15
* Candidate for systemic therapy or phototherapy in the opinion of the investigator
* Negative test for hepatitis B surface antigen, hepatitis C antibody, and Human Immunodeficiency Virus (HIV)
* Negative serum pregnancy test for female subjects (unless 3 years post menopausal or surgically sterile)
* Willing to use medically acceptable form of birth control for duration of study
* Negative Purified Protein Derivative (PPD) within 30 days prior to first dose of study drug

Exclusion Criteria:

* Any active infection
* Significant concurrent medical conditions, including: Insulin dependent diabetes mellitus; Congestive heart failure; Myocardial infarction within last year; Unstable angina pectoris; Uncontrolled hypertension; Severe pulmonary disease [requiring oxygen therapy or hospitalization]; Systemic lupus erythematosus; Multiple sclerosis or any other demyelinating disease; Active malignancy
* Any condition, in opinion of study doctor, that might cause this study to be detrimental to subject
* History of cancer within 5 years before first dose of study drug
* Skin conditions other than psoriasis that would interfere with evaluations of the effect of study medications on psoriasis
* Presence of guttate, erythrodermic or pustular psoriasis
* Use of topical cyclosporine or calcineurin inhibitors within 14 days of first dose of study drug
* Use of tar shampoos within 14 days of first dose of study drug
* Use of following therapies within 28 days of first dose of study drug: IV or oral cyclosporine or calcineurin inhibitors, Ultraviolet Light A therapy, Psoralen plus ultraviolet A radiation, Oral retinoids, Ultraviolet Light B therapy, Topical steroids or steroid shampoo, Topical vitamin A or D analog preparations, Anthralin, other systemic psoriasis therapy, cyclophosphamide, sulfasalazine, anakinra
* Use of Alefacept (Amevive), Efalizumab (Raptiva), Anti-tumor necrosis factor (TNF) biologic therapies within 3 months of the first dose of study drug. Prior anti-TNF use will not be permitted if discontinued due to lack of efficacy, an adverse event, or non-compliance.
* Use of interleukin (IL)-12/IL-23 within 6 months of the first dose of study drug
* Participation in another clinical trial within 90 days or 5 half-lives (whichever is longer) of randomization
* Laboratory abnormalities at screening: hemoglobin less than 11 g/dL, platelet count less than 125,000/mm^3, white blood cell count less than 3,500 cells/mm^3, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) greater than or equal to 1.5 x the upper limit of normal, any other laboratory abnormality which will prevent patient from completing the study or interfere with interpretation of study results
* Patient is pregnant or breast feeding
* Presence of any condition that could compromise the patient's ability to participate in the study, such as a history of substance abuse or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Bagel J, Lynde C, Tyring S, Kricorian G, Shi Y, Klekotka P. Moderate to severe plaque psoriasis with scalp involvement: a randomized, double-blind, placebo-controlled study of etanercept. J Am Acad Dermatol. 2012 Jul;67(1):86-92. doi: 10.1016/j.jaad.2011.07.034. Epub 2011 Oct 20. PMID 22014541
- [Background] Tyring S, Bagel J, Lynde C, Klekotka P, Thompson EH, Gandra SR, Shi Y, Kricorian G. Patient-reported outcomes in moderate-to-severe plaque psoriasis with scalp involvement: results from a randomized, double-blind, placebo-controlled study of etanercept. J Eur Acad Dermatol Venereol. 2013 Jan;27(1):125-8. doi: 10.1111/j.1468-3083.2011.04394.x. Epub 2011 Dec 21. No abstract available. PMID 22188302
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 5 December 2008 through 6 January 2010
Period: Weeks 1 to 12
Arm/Group | Placebo BIW/Etanercept 50 mg BIW | Etanercept 50 mg BIW/Etanercept 50 mg QW
Started | 62 | 62
Treated | 62 | 59
Completed | 54 | 58
Not Completed | 8 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Disease progression | 3 | 0
Not completed — Ineligibility determined | 0 | 3
Period: Weeks 13 to 24
Arm/Group | Placebo BIW/Etanercept 50 mg BIW | Etanercept 50 mg BIW/Etanercept 50 mg QW
Started | 54 | 57 (1 participant discontinued due to an adverse event after completing 12 weeks.)
Completed | 49 | 49
Not Completed | 5 | 8
Not completed — Protocol deviation | 2 | 0
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Disease progression | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BIW/Etanercept 50 mg BIW | Etanercept 50 mg BIW/Etanercept 50 mg QW | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.68 (13.79) | 41.55 (13.93) | 42.11 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 36 | 33 | 69
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 47 | 43 | 90
  Black or African American | 6 | 5 | 11
  Hispanic or Latino | 6 | 8 | 14
  Asian | 2 | 3 | 5
  American Indian or Alaska Native | 0 | 1 | 1
  Aborigine | 0 | 1 | 1
  Other | 1 | 1 | 2
Body Mass Index Group [Number; unit: participants]
  ≤ 35 kg/m^2 | 46 | 44 | 90
  > 35 kg/m^2 | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Psoriasis Scalp Severity Index at Week 12
Description: The Psoriasis Scalp Severity Index (PSSI) measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored by physicians using a scale from 0 to 72, where 0 = no psoriasis, and higher scores indicating more severe disease. The PSSI calculation does not include the face or neck area.
Time Frame: Baseline and Week 12
Population: Intention-to-Treat population (all patients who were randomized to investigational product) with available data; last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo BIW/Etanercept 50 mg BIW | Etanercept 50 mg BIW/Etanercept 50 mg QW
Number analyzed (Participants) | 61 | 59
Percent change | 20.4 (5.0) | 86.8 (2.3)
Statistical Analysis 1: Comparison: Placebo BIW/Etanercept 50 mg BIW vs Etanercept 50 mg BIW/Etanercept 50 mg QW; Test type: Superiority or Other; p < 0.0001, van Elteren's test; Stratified by baseline body mass index group

2. Secondary Outcome: Percentage of Participants With PSSI 75% Response at Week 12
Description: Percentage of participants achieving at least a 75% improvement from baseline in the Psoriasis Scalp Severity Index (PSSI) at Week 12. The Psoriasis Scalp Severity Index (PSSI) measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored by physicians using a scale from 0 to 72, where 0 = no psoriasis, and higher scores indicating more severe disease. The PSSI calculation does not include the face or neck area. PSSI 75 indicates at least a 75% improvement in the PSSI score from baseline.
Time Frame: Baseline and Week 12
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo BIW/Etanercept 50 mg BIW | Etanercept 50 mg BIW/Etanercept 50 mg QW
Number analyzed (Participants) | 61 | 59
Percentage of participants | 11 | 86
Statistical Analysis 1: Comparison: Placebo BIW/Etanercept 50 mg BIW vs Etanercept 50 mg BIW/Etanercept 50 mg QW; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by baseline body mass index group

3. Secondary Outcome: Percent Change From Baseline in PSSI at Week 24 in Participants Switching From Placebo to Etanercept at Week 12
Description: Percent change from baseline in Psoriasis Scalp Severity Index (PSSI) in participants switching from placebo to etanercept at Week 12 (Group B) at Week 24. The PSSI measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored by physicians using a scale from 0 to 72, where 0 = no psoriasis, and higher scores indicate more severe disease. The PSSI calculation does not include the face or neck area.
Time Frame: Baseline and Week 24
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo BIW/Etanercept 50 mg BIW
Number analyzed (Participants) | 61
Percent change | 79.1 (4.3)
Statistical Analysis 1: Comparison: Placebo BIW/Etanercept 50 mg BIW; Comparison of week 24 outcome to week 12 outcome (see Outcome Measure 1); Test type: Superiority or Other; p < 0.0001, 2-sided pairwise van Elteren's test; Stratified by baseline body mass index group

4. Secondary Outcome: Patient Satisfaction With Treatment at Week 12
Description: This response scale was adapted from the Medical Outcomes Study: Patient Satisfaction Survey. To assess satisfaction with treatment, the participant was asked to check a box (from "very dissatisfied" to "very satisfied") to indicate his or her level of satisfaction with the medication's control of psoriasis.
Time Frame: 12 Weeks
Population: Intention-to-Treat with available data at week 12; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: participants
Arm/Group | Placebo BIW/Etanercept 50 mg BIW | Etanercept 50 mg BIW/Etanercept 50 mg QW
Number analyzed (Participants) | 59 | 58
participants
  Very dissatisfied | 15 | 9
  Dissatisfied | 20 | 1
  Neither satisfied nor dissatisfied | 13 | 4
  Satisfied | 5 | 17
  Very satisfied | 6 | 27
Statistical Analysis 1: Comparison: Placebo BIW/Etanercept 50 mg BIW vs Etanercept 50 mg BIW/Etanercept 50 mg QW; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Two-sided test with modified ridit scores stratified by baseline body mass index group

ADVERSE EVENTS:
Time Frame: First dose to last dose +30 days (up to 28 weeks)
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo BIW/Etanercept 50 mg BIW | Etanercept 50 mg BIW/Etanercept 50 mg QW
Serious Adverse Events (participants affected / at risk) | 1/62 | 2/59
Other Adverse Events (participants affected / at risk) | 25/62 | 27/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BIW/Etanercept 50 mg BIW (N=62) | Etanercept 50 mg BIW/Etanercept 50 mg QW (N=59)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BIW/Etanercept 50 mg BIW (N=62) | Etanercept 50 mg BIW/Etanercept 50 mg QW (N=59)
INJECTION SITE REACTION (General disorders) | 3 | 4
BRONCHITIS (Infections and infestations) | 2 | 3
EAR INFECTION (Infections and infestations) | 4 | 0
NASOPHARYNGITIS (Infections and infestations) | 5 | 5
SINUSITIS (Infections and infestations) | 1 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 4
HEADACHE (Nervous system disorders) | 2 | 4
HYPERTENSION (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.